CLINICAL TRIAL: NCT05433792
Title: An Open Label, 3 Arms, Multicenter, Randomized . To Evaluate the Effectiveness Fitlens Soft Central Near and Central Far Contact Lens, Compared With MiSight for the Control of Progressive Juvenile Onset Myopia in Children Ages 8-12.
Brief Title: To Evaluate the Effectiveness of New Specially Designed Fitlens Soft Lens.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fitlens Ltd. (Industry)
Collaborators: RSNESS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FL-CN/CF-01
Record Dates: First submitted 2022-06-07; First posted 2022-06-27 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Intervention Model Description: This is an open label, 3 arms, Multicenter, randomized study to evaluate the effectiveness of new specially designed Fitlens soft central near and central far contact lens, Myolens CN/CF Compared with MiSight® for the control of progressive juvenile onset Myopia in children ages 8-12. with no prior contact lens experience. Subjects will be allocated to either of the study arms - CN / CF or MiSight in a 1:1:1 ratio. The randomization for each arm will be done regardless the Myopia categories.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Myolens CN (Experimental): Subjects' will be allocated to Myolens CN study arm in a 1:1:1 ratio.
  Interventions: Device: Myolens CN (Central-Near) soft contact lens
- Myolens CF (Experimental): Subjects' will be allocated to Myolens CF study arm in a 1:1:1 ratio.
  Interventions: Device: Myolens CN (Central-Near) soft contact lens
- MiSight® (Active Comparator): Subjects' will be allocated to MiSight® study arm in a 1:1:1 ratio.
  Interventions: Device: MiSight® soft contact lens

INTERVENTIONS:
Device: Myolens CN (Central-Near) soft contact lens — Personal fitting of the Myolens-CN/CF.
  Other Names: Myolens CF (Central-Far) soft contact lens
  Arms: Myolens CF; Myolens CN
Device: MiSight® soft contact lens — Control arm device, FDA approved (P180035), and CE marked soft lenses for the management of Myopia in children aged 8-12.
  Arms: MiSight®

SUMMARY:
Myopia is a common disorder, affecting approximately one-third of the US population and over 90% of the population in some East Asian countries. High amounts of myopia are associated with an increased risk of sight-threatening problems, such as retinal detachment, choroidal degeneration, cataracts, and glaucoma. Slowing the progression of myopia could potentially benefit millions of children. To date, few strategies used for myopia control have proven to be effective. Currently, there are four categories of myopia control treatments: atropine eye drops, multifocal contact lenses, multifocal eyeglasses, and orthokeratology (ortho-k). None of these modalities are US Food and Drug Administration-approved to slow myopia progression, they have been shown to slow the progression by approximately 50% with few risks. Both orthokeratology and soft bifocal contact lenses have shown to slow myopia progression by slightly less than 50% in most studies.

The Myolens progressive front soft contact lens is designed to slow down myopia progression in children, The Myolens lens is an aspheric design with a spherical back surface that provides clear vision, with a uniform round edge for excellent fit and optimum comfort.

The Myolens-CN is designed with a central for the near optics, while the Myolens-CF with a central for the distance optics, which progressively changes to far area and within a defined optical zone area while considering the movement up-down of the lens on the cornea.

The thought behind the design is that the center of the lens will not provide a full optical correction.

In the suggested study, both Myolens modalities CN and CF will be investigated in compare to the current approved treatment - MiSight.

DETAILED DESCRIPTION:
Study Procedures:

Screening period (up to 3 weeks prior to enrollment)

1. Obtaining inform consent.
2. Obtaining subject's relevant medical history and concomitant therapy - concurrent active medical conditions with emphasis on ocular and systemic diseases.
3. Performance of ophthalmic examination (slit lamp), IOP, BCVA, cycloplegia refractive, axial length measurement, spherical equivalent calculation, Cover test, fundus photography and corneal topography.
4. Confirmatiom of subject's eligiblity
5. Subject's randomization to either of the study arms
6. Personal fitting of the Myolens-CN/CF or MiSight as per randomization

Week 1 Day 1 (±3 days)

1. Performance of ophthalmic examination (slit lamp), BCVA, cycloplegia refractive, axial length measurement, spherical equivalent calculation.
2. Subject will be instructed regarding the use and handling of the lens both written and verbally.
3. AE and concomitant therapy monitoring

Treatment period (36 months)

1. The lenses will be worn by the subject every day, for a maximum of 14 hours per day.
2. For the subjects allocated to either CN or CF arm, lenses will be replaced every 3 months.
3. At M36 visit lenses will be removed.
4. Each follow up visit will include: ophthalmic examination (slit lamp), BCVA test , axial length measurement, refractive assessment and spherical equivalence calculation, subject diary review, AE monitoring and changes in concomitant medications.

Follow up period (4 weeks) End of study (EOS) visit will be conducted 4 weeks after EOT. Completion of the study will be considered as the completion of visit 36M which will the EOT visit for the subject and 4 weeks follow up. In case of early termination, EOS will be conducted upon time of termination (UNS). EOS visit procedures are equal to 36M visit procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Be between 8 and 12 years of age inclusive at baseline examination.
2. The participant has been given a detailed, clear explanation concerning the study aspects and procedures.
3. The participant's parents or legal guardian have been given a clear explanation, then read, understood, and signed the informed consent form.
4. Willingness to adhere to protocol, agreement to maintain the visit schedule.
5. Along with their parent or guardian, agree to maintain the visit schedule and be able to keep all appointments as specified in the study protocol for the duration of the study.
6. Agreement to wear the assigned contact lenses for a minimum of 10 hours per day, at least 6 days per week, for the duration of the 3-year study.
7. Subject with normal eyes who is not using any ocular medications.
8. Possess wearable and visually functional eyeglasses.
9. Be in good general health, based on his/her and parent's/guardian's knowledge.
10. Best-corrected visual acuity by manifest refraction of +0.10 log MAR (20/25 or 6/7.5) or better in each eye. (Lens power required limited to up to minus 10).
11. The manifest cylinder is less than or equal to 0,75D.
12. Meet the following refractive criteria determined by cycloplegic autorefraction at baseline (per eye):

    1. Spherical equivalent refractive error: between -0.75 and -4.00 D inclusive.
    2. Astigmatism: ≤-0.75 D
    3. Anisometropia: <1.00 D

Exclusion Criteria:

1. Subject is currently or within 30 days before this study has been an active participant in another clinical study involving an investigational treatment.
2. Current or prior use of bifocals, progressive addition lenses, atropine, pirenzepine, or any other myopia control treatment.
3. Birth earlier than 30 week or <1500 g (3.3 lb) at birth.
4. Regular use of ocular medications, artificial tears, or wetting agents.
5. Current use of systemic medications, which may affect contact lens wear, tear film production, pupil size, accommodation, or refractive state.
6. A known allergy to any of the Myolens components.
7. A history of corneal hypoesthesia (reduced corneal sensitivity), corneal ulcer, corneal infiltrates, ocular viral or fungal infections, or other recurrent ocular infections.
8. Strabismus by cover test at distance or near wearing distance correction.
9. History of any of the following: ocular or systemic diseases, including those that could influence refractive development, anterior segment infection, inflammation or abnormality, any active anterior segment ocular disease that would contraindicate contact lens wear; history of herpetic keratitis; history of refractive surgery or irregular cornea (except when the contact lenses under investigation are indicated for irregular cornea, keratoconus or refractive surgery); a pathologically dry eye.
10. Keratoconus or an irregular cornea (assessed by corneas topography)
11. Contraindications for contact lens wear including giant papillary conjunctivitis of grade 2 or worse and allergic or seasonal conjunctivitis (assessed by slit lamp exam)
12. Subject seems to exhibit poor personal hygiene (that in the investigator's opinion might prevent safe contact lens wear) or the investigator for any reason considers that it is not in the best interest of the subject to participate in the study.
13. Slit lamp findings that are more serious than grade 1 according to the Efron Grading Scale.
14. Corneal vascularization greater than 1 mm of penetration

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Axial length change from baseline visit to 12 months visit. | from baseline visit to 12 months visit
  Axial length change from baseline visit to 12 months visit.
Spherical equivalent change from baseline visit to 12 months visit. | from baseline visit to 12 months visit
  Spherical equivalent change from baseline visit to 12 months visit.

SECONDARY OUTCOMES:
BCVA change from baseline visit to 12 months visit. | from baseline visit to 12 months visit
  BCVA change from baseline visit to 12 months visit.
Axial length change from baseline visit to 24 months visit. | from baseline visit to 24 months visit
  Axial length change from baseline visit to 24 months visit.
Spherical equivalent change from baseline visit to 24 months visit. | from baseline visit to 24 months visit
  Spherical equivalent change from baseline visit to 24 months visit.
BCVA change from baseline visit to 24 months visit. | from baseline visit to 24 months visit
  BCVA change from baseline visit to 24 months visit.
Axial length change from baseline visit to 36 months visit. | from baseline visit to 36 months visit
  Axial length change from baseline visit to 36 months visit.
Spherical equivalent change from baseline visit to 36 months visit. | from baseline visit to 36 months visit
  Spherical equivalent change from baseline visit to 36 months visit.
BCVA change from baseline visit to 36 months visit. | from baseline visit to 36 months visit
  BCVA change from baseline visit to 36 months visit.
Axial length change in CN arm | Up to 36 months after last patient recruitment) = last subject enrolled study completion).
  Axial length change in CN arm
Spherical equivalent change in CN arm | Up to 36 months after last patient recruitment) = last subject enrolled study completion).
  Spherical equivalent change in CN arm
BCVA change in CN arm | Up to 36 months after last patient recruitment) = last subject enrolled study completion).
  BCVA change in CN arm
Axial length change in CF arm | Up to 36 months after last patient recruitment) = last subject enrolled study completion).
  Axial length change in CF arm
Spherical equivalent change in CF arm | Up to 36 months after last patient recruitment) = last subject enrolled study completion).
  Spherical equivalent change in CF arm
BCVA change in CF arm | Up to 36 months after last patient recruitment) = last subject enrolled study completion).
  BCVA change in CF arm

OTHER OUTCOMES:
Rate of device related Adverse Events. | Up to 36 months after last patient recruitment) = last subject enrolled study completion).
  Rate of device related Adverse Events.
Exploratory Endpoint. | Up to 36 months after last patient recruitment) = last subject enrolled study completion).
  Comparing CN and CF in change in axial length, spherical equivalate and BCVA.
Exploratory Endpoint. | Up to 36 months after last patient recruitment) = last subject enrolled study completion).
  Comparing CN and CF in change in spherical equivalate
Exploratory Endpoint. | Up to 36 months after last patient recruitment) = last subject enrolled study completion).
  Comparing CN and CF in change in BCVA.

CONTACTS AND LOCATIONS:
Overall Officials: Nitza Cohen, MD, Principal Investigator — Bnei- Zion MC. Israel; Oriel Shpirer, MD, Principal Investigator — Wolfson MC. Israel; Shiri Shulman, MD, Principal Investigator — Assuta- Hashalom MC. Israel; José M González Méijome, MD, Principal Investigator — University of Minho- Portugal
Locations (1):
- Wolfson Medical Center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No